CLINICAL TRIAL: NCT07082491
Title: Effectiveness of Mindfulness-Based Protocols in Reducing Work-Related Stress
Brief Title: Mindfulness for Reducing Work-Related Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: University of Siena, Italy (Unknown)
Responsible Party: Principal Investigator, Teresa Fazia, Principal Investigato, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mindfulness_Siena
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Work-Related Stress; Well-being; Inflammation Status; Employees of University
Keywords: mindfulness; stress; inflammation; biomarkers; employees of university; MBSR
MeSH Terms: conditions — Occupational Stress; Inflammation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The study involves two groups: one receiving the mindfulness-based intervention and a control group (waiting-list control). Participants are randomized into these two groups and followed in parallel without switching between conditions. The outcomes are measured before and after the intervention, comparing the effects between the two groups. Data were also collected at follow-up (1 month).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction (Experimental): Participants in this group will undergo a MBSR intervention. The intervention consists of 8 in-person sessions over 8 weeks, with each session lasting about three hours, once per week.
  Interventions: Behavioral: Mindfulness-based stress reduction
- Waiting-List Control Group (No Intervention): Participants in this group will not receive any intervention during the study period. They will be placed on a waiting list and instructed to refrain from any meditation or mindfulness-based activities until the study is completed. This group serves as a passive control to evaluate the effectiveness of our intervention by comparing pre- and post-intervention measures.

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — The intervention consists of 8 in-person sessions over a period of 8 weeks, with each session lasting about three hours, once per week, with an intensive full-day practice session lasting 7 hours. The instructors provide audio recordings at each session to be used as daily practice. The MBSR program is an introductory pathway to mindfulness practices that works through the systematic and continuous cultivation of specific mental states that foster a different relationship with stress.
  Arms: Mindfulness-based stress reduction

SUMMARY:
Work-related stress is a major contributor to absenteeism and reduces work productivity. Long-term chronic stress also has a detrimental impact on health and increases the risk of mental and physical illnesses. This underscores the urgency and need to find new approaches for the prevention and management of stress. Literature studies show that Mindfulness is an innovative and effective tool for managing stress in a variety of medical, social, and educational contexts. Mindfulness can be defined as a specific form of attention focused on the present moment, intentional and non-judgmental. Growing scientific evidence supports both the use and implementation of Mindfulness-Based Interventions (MBIs) in workplace settings to improve the ability to manage work-related stress and to enhance resilience. However, despite the increasing popularity and diffusion of MBIs, the biological mechanisms underlying the beneficial effects of Mindfulness remain unclear.

The present study aims to evaluate the effectiveness of a Mindfulness-Based Stress Reduction (MBSR) program in improving physical and psychological well-being in a workplace setting (University of Siena). Specifically, this study will assess the impact of MBSR on stress reduction using an intervention adapted to the specific needs and requirements of the workplace.

Additionally, the investigators will investigate whether MBSR can influence psychological correlates and biological markers of stress (inflammatory markers) in these employees. The effectiveness of this intervention could lead to an improvement in employees' quality of life and health and to a reduction in the socioeconomic impact of stress.

DETAILED DESCRIPTION:
Chronic stress has been associated with conditions such as diabetes (Hilliard et al., 2016), gastrointestinal diseases (Mayer, 2000), metabolic syndrome (Chandola et al., 2006), hyperthyroidism (Tsigos and Chrousos, 2002), cardiovascular diseases (Rosengren et al., 2004) and strokes caused by stressful work conditions (Huang et al., 2015). Strong experimental evidence shows the involvement of stress in mental disorders such as depression (Slavich and Irwin, 2014) and anxiety (O'Donovan et al., 2013). An individual exposed to intense and prolonged stress stimuli may experience cognitive disorders: the person has greater difficulty maintaining concentration, loses interest in work and other usual activities (hobbies, sports), and undergoes mood changes (depression, anxiety, emotional detachment, etc.). Changes are also observed in behavior, including eating disorders (such as anorexia nervosa or bulimia), and in more severe cases, obsessive-compulsive disorders (Tsigos and Chrousos, 2002).

The current regulatory framework for health and safety in the workplace has identified work-related stress as one of the main risks to the physical and mental well-being of workers. The European Commission [report by the European Agency For Safety and Health at Work (2009), European Foundation For the Improvement of Living and Working Condition (2006)] reports that work-related stress affects 22% of European workers and 27% of Italian workers. Studies carried out by the European Commission in 2002 also showed the relative economic cost of work-related stress, suggesting that 50-60% of lost workdays are due to stress, with an annual economic cost of 20 billion euros. Investing in programs that help manage and reduce work-related stress, increasing well-being, can therefore help reduce these costs and increase company productivity.

Among the practices proposed to increase resilience and improve stress management, including in the workplace, Mindfulness is an innovative and particularly effective tool. Mindfulness can be defined as a specific form of attention that is (1) focused on the present moment, (2) intentional, and (3) non-judgmental (Kabat-Zinn, 2005). Mindfulness-Based Interventions (MBIs) offer mental training that enhances our capacity for attention, concentration, and calm, developing an attitude of awareness, curiosity, openness, and acceptance of all the experiences, including negative ones. In these interventions, participants intensively practice awareness both during group sessions and through daily tasks. Moreover, practice instructions are integrated with psycho-educational content to address stress, anxiety, or depressive symptoms.

MBIs (in particular the Mindfulness-Based Stress Reduction program - MBSR) have proven effective in managing stressful events in the workplace (Hulsheger et al., 2013; Koncz et al., 2016). In recent years, MBIs have attracted the attention of industrial and organizational psychology scholars as a means to reduce workplace stress and improve employee engagement and productivity. Preliminary evidence shows positive effects on empowerment and engagement, as well as on burnout, in physicians. Their effectiveness has also been demonstrated in reducing emotional exhaustion and improving sleep quality in workers. Studies in the business field indicate that MBIs are beneficial for improving service quality, and performance levels in various tasks. Today, many large companies (such as Apple, Google, Nike, Procter & Gamble, Deutsche Bank, General Mills, etc.) or business schools have recognized the benefits of Mindfulness in organizations and offer MBIs to their managers, employees, and students.

Despite its growing popularity, the neurobiological mechanisms underlying the health benefits of Mindfulness are still poorly understood. In a previous study, it was reported a significant increase in the thickness of the insula and somatosensory cortex in university students who completed an 8-week Mindfulness program. These areas are associated with interoception, body movement awareness, and emotional awareness. These changes were associated with a reduction in psychological indices such as worry, anxiety, and depression. Mindfulness practice, by training interoception, can improve the understanding and processing of emotional reactions to internal and external stimuli, decreasing reactivity and improving stress response.

Although many studies show that MBIs can improve symptoms related to stress, the biological mechanisms underlying the beneficial effect of Mindfulness are still not well understood. For this reason, in a preliminary study conducted on healthy subjects, it was evaluated the effect of intensive Mindfulness practice (3-day intensive) on psychological and biological parameters associated with stress (Gardi et al. Changes in salivary cytokine production in subjects attending a 3-day mindfulness retreat: a pilot study. "Second International Conference on Mindfulness", Rome 2016; Gardi C. et al. manuscript in preparation). The Mindfulness group was compared with an active control group, matched for age and sex. The intensive training significantly reduced salivary cortisol levels (the main stress hormone) and some inflammatory markers (such as IL-6 and IL-8). In the Mindfulness group, an increase in awareness and a decrease in perceived stress and anxiety were also observed. The described study is the first to document significant correlations between intensive Mindfulness practice and positive psychological changes, together with inflammatory status. These results, although preliminary, suggest that Mindfulness practice can not only help alleviate psychological distress but also contribute to improving certain inflammation biomarkers, with important implications for health.

In this project, the investigators propose a MBSR intervention which may have significant implications for employee health, their performance, and a reduction in company costs.

The present study aims to evaluate the effectiveness of this intervention in improving physical and psychological well-being in a workplace context (University of Siena). Specifically, the investigators will assess the impact of Mindfulness practice on stress reduction using an intervention tailored to the specific needs and requirements of the workplace.

Additionally, the investigators will investigate whether Mindfulness training can influence psychological correlates and biological markers of stress (inflammatory and oxidative markers) in these employees. The effectiveness of this intervention could lead to an improvement in employees' quality of life and health and to a reduction in the socioeconomic impact of stress.

Primary Endpoint: Improvement in scores from questionnaires measuring distress, burnout, and, in parallel, an increase in psychological well-being and self-awareness.

Secondary Endpoints: Reduction in stress- and inflammation-related markers (i.e., cortisol, cytokines).

Stabilization of the changes observed in participants at the end of the treatment (1-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Employees of the University of Siena who agree (and are motivated) to participate in the Mindfulness protocol, aged over 18 years and ≤ 65 years.
* Willingness to provide free and informed consent.

Exclusion Criteria:

* Use of psychotropic medication in the last 2 months
* Unwillingness to sign the informed consent form
* Medical conditions that prevent participation in group sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Reduction in distress and burnout as measured by the Perceived Stress Scale (PSS) and Maslach burnout inventory (MBI) | Baseline (T0), post-intervention (8 weeks, T1), follow-up (1 month, T2)
  The mprovements in scores from PSS and MBI questionnaire measuring distress and burnout, indicate enhanced psychological well-being and decreased vulnerability to chronic stress.

SECONDARY OUTCOMES:
Improvmente in present-moment attention and awareness, as measured by the Mindful Attention Awareness Scale (MAAS) | Baseline (T0), post-intervention (8 weeks, T1), follow-up (1 month, T2)
  The improvement in MAAS scores reflects enhanced moment-to-moment self-awareness and greater attentional engagement in daily experiences
Reduction of anxiety as measured by State anxiety inventory (STAI) | Baseline (T0), post-intervention (8 weeks, T1), follow-up (1 month, T2)
  The decrease in STAI scores reflects a significant reduction in anxiety levels, indicating improved emotional regulation and lower acute stress in response to contextual demands.
Reduction in stress biomarker measured in saliva sample | Baseline (T0), post-intervention (8 weeks, T1), follow-up (1 month, T2)
  Cortisol was assayed using standard enzyme-linked immunoassay procedures . Samples were assayed in duplicate and averaged. Lower limit of detection was 0.07 ng/ml; intra and inter-assay variation had coefficients of covariance at less than 10%. Reduction in cortisol levels indicates a decreased physiological stress response
Reduction in inflammation-related markers measured in saliva sample | Baseline (T0), post-intervention (8 weeks, T1), follow-up (1 month, T2)
  Salivary concentrations of cytokines (IL-6 and IL-8) were measured according to manufacturer specifications using the Bio-Plex Pro Assays. Bio-Plex Pro Assays are immunoassays formatted on magnetic beads that utilize principles similar to those of a sandwich ELISA. Capture antibodies against the biomarker of interest are covalently coupled to the beads. A biotinylated detection antibody creates the sandwich complex, and the final detection complex is formed by the addition of a streptavidin-phycoerythrin (SA-PE) conjugate, where PE serves as the fluorescent reporter. Reactions are read using a Luminex-based reader. All assays were performed in duplicate to maximize reliability. Reduction in IL-6 and IL-8 levels indicates a decrease in systemic inflammation and immune activation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Siena, Siena, Italy